CLINICAL TRIAL: NCT02762292
Title: Work of Breathing Assessment During Weaning From Mechanical Ventilation
Acronym: WOAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, MD PHD, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUSJ 2017-1259
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Mechanical Ventilation
Keywords: Mechanical ventilation; Children; Work of breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental)
  Interventions: Device: Measurement of work of breathing using indirect calorimeter

INTERVENTIONS:
Device: Measurement of work of breathing using indirect calorimeter — 1. Preparation:
     1. Patient baseline characteristics will be collected.
     2. Connection of the Indirect Calorimeter to the respiratory circuit.
     3. Nasogastric tube installation: a specific modified Neurally Adjusted Ventilatory Assist (NAVA) catheter equipped with both microelectrodes for Electrical Activity of the diaphragme (EAdi) monitoring and an esophageal balloon (for esophageal pressure (PES) monitoring) will be installed.
  2. Simultaneous recordings of: Oxygen Consumption (VO2) and Energy Expenditure (EE); Esophageal Pressure (PES), Airway Pressure (PAW), respiratory volume and flow; EAdi during (i) Conventional mechanical ventilation (ii) Spontaneous Breathing Trial in Continuous Positive Airway Pressure and (iii) Second period of Conventional mechanical ventilation with the same ventilator parameters set in STEP 1.
  3. End of the physiological recordings. Collection of Pediatric Intensive Care Unit (PICU) outcome of patients.

SUMMARY:
Introduction In patients assisted by mechanical ventilation, the Work Of Breathing (WOB) is shared between the patient and the ventilator. During weaning from mechanical ventilation, the WOB performed by the patient must be adequate and efficient to sustain spontaneous ventilation after extubation. The monitoring of WOB during weaning might allow a better management of the weaning process. Esophageal pressure (PES) is the reference technique to measure WOB but alternate tools have been proposed. The main hypothesis is that Indirect Calorimetry (IC) is valid to track the changes in energy expenditure due to the changes in WOB in mechanically ventilated children during weaning from mechanical ventilation. The primary objective of this study is to assess the validity of IC method for the WOB assessment when compared to PES measurement and Electrical Activity of the diaphragm (EAdi) during a spontaneous breathing trial (SBT) in continuous positive airway pressure, which is a routine extubation readiness test which generally induces an increase in WOB.

Methods This is a prospective single center study. All intubated and mechanically ventilated children >1 months and <18 years old, hospitalized in the pediatric intensive care unit will be eligible.

Simultaneous recordings of Energy Expenditure, PES and EAdi will be performed during 3 steps: before, during and after the SBT. Then outcome of patients will be collected.

The investigators plan to study a sample of 15 patients to be representative.

Relevance to the importance of child health in Canada The investigators expect that the IC-based less invasive method will provide an accurate estimation of WOB assessment. Once this tool is validated, the interest of IC to (i) early detect an increase in WOB during mechanical ventilation in children, (ii) to assess the ability to extubate them and (iii) to optimize nutritional support will be assessed in future studies.

ELIGIBILITY:
Inclusion Criteria:

All intubated and mechanically ventilated children >1 months and <18 years old, hospitalized in the pediatric intensive care unit will be eligible.

The patient is deemed to be ready for an extubation readiness test as per the attending team. In particular, the following criteria should be met:

* Improvement in the underlying condition that led to intubation;
* Presence of spontaneous breathing, and adequate oxygenation:, FiO2 ≤ 0.6 (to obtain a SpO2 between 92 and 97%), with Positive End Expiratory Pressure < 8 cmH2O;
* Adequate mental status: Arousal;
* Effective cough;
* No planned operative procedure requiring heavy sedation in the next 12 hours.

Exclusion Criteria:

* Contraindications to the placement of a new nasogastric tube (e.g. trauma or recent surgery in cervical, esophageal, or nasopharyngeal regions, severe coagulation disorder);
* Hemodynamic instability requiring milrinone ≥ 0.5µg/kg/min, dopamine ≥ 5µg/kg/min, epinephrine ≥ 0.03µg/kg/min, norepinephrine ≥ 0.03µg/kg/min, or dobutamine ≥ 5µg/kg/min;
* Severe respiratory instability, and in particular PaCO2 > 80 mmHg on the last blood gas in the last 4 hours;
* Axillary temperature >38°;
* Cuff leaks >10%, calculated by the ventilator as mean inspired tidal volume minus mean expired tidal volume divided by inspired tidal volume;
* Absence of parental or tutor consent;
* Patient for whom a limitation of life support treatments is discussed or decided.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Consumption, measured during 3 periods of 30 minutes: before (STEP 1), during (STEP 2) and after (STEP 3) the SBT. | Up to 2 hours from the beginning of the study
Change in Energy Expenditure, measured during 3 periods of 30 minutes: before (STEP 1), during (STEP 2) and after (STEP 3) the SBT. | Up to 2 hours from the beginning of the study

SECONDARY OUTCOMES:
Change in Esophageal pressure | Up to 2 hours from the beginning of the study
  Esophageal, calculated as the mean value of 10 consecutive breaths, before (STEP 1), during (STEP 2) and after (STEP 3) the SBT;
Change in Esophageal pressure time product | Up to 2 hours from the beginning of the study
  Pressure Time Product, calculated as the mean value of 10 consecutive breaths, before (STEP 1), during (STEP 2) and after (STEP 3) the SBT;
Change in Electrical Activity of the diaphragm (EAdi) | Up to 2 hours from the beginning of the study
  EAdi, calculated as the mean inspiratory value during 1 minute, before (STEP 1), during (STEP 2) and after (STEP 3) the SBT;
Change in Respiratory Rate | Up to 2 hours from the beginning of the study
  Respiratory Rate, monitored during the SBT;
Change in Cardiac Rate | Up to 2 hours from the beginning of the study
  Cardiac Rate, monitored during the SBT;
Duration of mechanical ventilation | Up to 3 months
Spontaneous Breathing test success or failure | Up to 28 hours
  extubation success or failure (as defined by the need to re-intubate in the 24 hours following extubation).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada